CLINICAL TRIAL: NCT02426203
Title: Three-dimensional Echocardiographic Assessment of Right Ventricular Function in Patients Undergoing Pulmonary Endarterectomy
Brief Title: 3D Echocardiographic Assessment of RV Function in Patients Undergoing Pulmonary Endarterectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: P02016
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Echocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulmonary Endarterectomy patients: Patients undergoing pulmonary endarterectomy surgery at Papworth Hospital
  Interventions: Procedure: Pulmonary endarterectomy

INTERVENTIONS:
Procedure: Pulmonary endarterectomy — Echocardiographic assessment right ventricular function prior to, during, and following Pulmonary Endarterectomy surgery.
  Other Names: Transoesophageal Echocardiography; Transthoracic Echocardiography

SUMMARY:
Chronic thromboembolic pulmonary hypertension causes progressive right heart hypertrophy, dilatation and dysfunction. Surgical treatment is pulmonary endarterectomy, which although only carried out in a single UK centre, provides an excellent model for assessing right ventricular function. Right heart function is most commonly assessed using echocardiography, either transthoracic pre- and post-operatively, or transoesophageal intra-operatively. Measurement of tricuspid annular plane systolic excursion is the best validated and most commonly performed measurement for right heart function, however it may be inaccurate after sternotomy and pericardial opening, making accurate assessment difficult immediately after surgery. Therefore, we aim to compare established methods of assessing right heart function with 3-dimensional echocardiographic reconstruction of the ventricle, using a novel reconstruction mechanism. Right ventricular function will be assessed in 51 patients who undergo pulmonary endarterectomy surgery at baseline, after the pericardium has been opened, following the surgical procedure, using transoesophageal echocardiography, and at six-month outpatient followup using transthoracic echocardiography, as 3D-reconstruction is valid using both modalities. This comparison should allow the investigators to determine whether such a method could replace current measurement parameters for assessment of right ventricular function, which is important for clinical management of patients in a variety of settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* undergoing pulmonary endarterectomy surgery at Papworth Hospital
* Willing to provide informed consent

Exclusion Criteria:

* Patient refusal
* Contraindication to transoesophageal echocardiography
* Technical difficulty preventing adequate echocardiographic assessment of right heart function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic thromboembolic pulmonary hypertension who are undergoing pulmonary endarterectomy surgery
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Right ventricular ejection fraction | 6 months
  3-dimensional acquisition of right ventricular ejection fraction using echocardiography

SECONDARY OUTCOMES:
Tricuspid annular plane systolic excursion | 6 months
Right ventricular fractional area change | 6 months
Right ventricular strain | 6 months
Pulmonary artery acceleration time | 6 months
Left ventricular ejection fraction | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Roscoe, FRCA, Principal Investigator — Papworth Hospital NHS Foundation Trust